CLINICAL TRIAL: NCT05036564
Title: Mutational Analysis in the Cerebrospinal Fluid to Improve Diagnostic Sensitivity, Response Definition and Precision Treatment in Primary Central Nervous System Lymphoma
Brief Title: Diagnosis; Objective RespOnse; THErApy
Acronym: DOROTHEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Teresa Calimeri (Unknown); Sara Steffanoni (Unknown)
Responsible Party: Principal Investigator, Andrés José Maria Ferreri, Principal Investigator; Lymphoma Unit, Head, IRCCS San Raffaele
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DOROTHEA
Record Dates: First submitted 2021-05-07; First posted 2021-09-05 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Primary CNS Lymphoma
Keywords: PCNSL; ctDNA; CSF
MeSH Terms: interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study population - PCNSL (Experimental): Patients (pts) with clinical and radiological suspicion of PCNSL or with confirmed diagnosis of PCNSL will be enrolled to the protocol. They will represent the "Study population"
  Interventions: Procedure: Lumbar puncture
- Control (Other): 1. Pts with suspicion of secondary CNS lymphoma, that includes subjects with DLBCL and involvement of the CNS at presentation in association with systemic disease, or subjects with systemic DLBCL and CNS relapse during or after primary therapy.
  2. Pts with histological diagnosis of systemic DLBCL at high risk of CNS relapse according to Institutional guidelines and patients with histological diagnosis of systemic high grade B cell lymphoma, according to 2017 WHO classification;
  3. pts affected by neurological disorders that are usually differential diagnosis of PCNSL (i.e. neurodegenerative and neuroinflammatory disorders, toxic or infective encephalitis, other primary CNS tumors).
  Interventions: Procedure: Lumbar puncture

INTERVENTIONS:
Procedure: Lumbar puncture — A lumbar puncture (spinal tap) is performed in patient lower back, in the lumbar region.
  During a lumbar puncture, a needle is inserted between two lumbar bones (vertebrae) to remove a sample of cerebrospinal fluid (CSF). This is the fluid that surrounds brain and spinal cord to protect them from injury.
  This procedure is usually performed at the time of diagnosis for disease staging and/or repeated in the course of the disease history, only if positive or for clinical reasons (i.e. suspicious of relapse progression).
  In this study sequential CSF and peripheral blood samples of study population will be collected also at different time points, with the aim to improve diagnostics sensitivity, response assessment and monitoring early CNS relapse.

SUMMARY:
Thi is a prospective and low-intervention clinical trial. We propose to design a panel of "core" genetic alterations by sequencing Cerebral Spinal Fluid (CSF) DNA in patients with confirmed or suspicious Primary Central Neurvous System Lymphoma (PCNSL) with the aim to improve diagnostic sensitivity, response assessment and monitoring early CNS relapse in routine practice.

Enrolled patients will receive conventional treatments according to well-established international guidelines, DNA assessments will not influence the treatment choices.

ELIGIBILITY:
Inclusion Criteria for study population:

1. Age ≥18 years
2. Newly diagnosed PCNSL with available clinical and radiological data, CSF and histopathological brain biopsy material fresh and/or formalin fixed and paraffin embedded;
3. No contraindications to stereotactic or open brain biopsy and lumbar puncture;
4. No formal contraindications to intravenous chemo-immunotherapy or whole-brain irradiation;
5. Given written informed consent prior to any study specific procedures, with the understanding that the patient has the right to withdraw from the study at any time, without any prejudice.

Exclusion Criteria for study population:

1. Patients with concomitant CNS and systemic involvement at presentation (potentially eligible as "control"; see below)
2. Patients with CNS lymphoma other than DLBCL subtype
3. Any other serious medical condition which could impair the ability of the patient to participate in the trial
4. Pregnant and lactating female patients. Sexually active patients of childbearing potential must implement adequate contraceptive measures during study participation.
5. Previous or concurrent malignancies at other sites diagnosed or relapsed within the last 3 years before PCNSL diagnosis. Patients with surgically cured in situ carcinomas and basal cell carcinoma of the skin are allowed.
6. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Inclusion criteria for controls:

1. Age ≥18 years
2. Newly diagnosed DLBCL with a high risk for relapse/progression in the CNS or High-grade B-cell (HGBC) lymphoma with available clinical and radiological data, CSF and diagnostic histopathological specimen. 3. Newly diagnosed and/or relapsed SCNSL with available clinical and radiological data, CSF and diagnostic histopathological specimen. 4. Newly diagnosed lymphoma confined to CNS other than DLBC subtype 5. Neoplastic and non-neoplastic neurological disorders (neurodegenerative and neuroinflammatory disorders, toxic or infective encephalitis, primary CNS tumors other than lymphomas (mainly gliomas)) with available clinical and radiological data, CSF samples and, where possible, histo-pathological brain biopsy material formalin fixed and paraffin embedded.

6. No contraindications to stereotactic or open brain biopsy and lumbar puncture; 7. Given written informed consent prior to any study specific procedures, with the understanding that the patient has the right to withdraw from the study at any time, without any prejudice.

Exclusion criteria for controls:

1. Patients with extra-CNS lymphoma other than DLBC or HGBC subtypes, and not classified as high risk of CNS relapse;
2. Any other serious medical condition which could impair the ability of the patient to participate in the trial;
3. Pregnant and lactating female patients. Sexually active patients of childbearing potential must implement adequate contraceptive measures during study participation;
4. Previous or concurrent malignancies at other sites diagnosed or relapsed within the last 3 years of follow-up. Patients with surgically cured in situ carcinomas and basal cell carcinoma of the skin are allowed;
5. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-10-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Association between recurrent genetic alterations and PCNSL diagnosis or relapse | 3 years and 6 months
  Frequency of various genetic mutations among enrolled patients at diagnosis or relapse
Association between recurrent genetic alterations and residual enhanced and not-enhanced images at the MRI | 3 years and 6 months
  Frequency of various genetic mutations among enrolled patients during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrés J.M. Ferreri, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy/Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No